CLINICAL TRIAL: NCT00925769
Title: An Open Label Study to Evaluate the Safety and Effect on Disease Progression of Triple Combination Treatment With Erlotinib (Tarceva), Bevacizumab (Avastin), and Capecitabine (Xeloda) in Patients With Locally Advanced and/or Metastatic Pancreatic Cancer (REBECA-Trial).
Brief Title: ATX Study:A Study of Avastin (Bevacizumab), Tarceva (Erlotinib) and Xeloda (Capecitabine) in Patients With Locally Advanced and/or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20784; 2008-004444-36
Record Dates: First submitted 2009-04-15; First posted 2009-06-22 (Estimated); Results first posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Capecitabine; Erlotinib Hydrochloride

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: capecitabine [Xeloda]; Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: bevacizumab [Avastin] — Escalating doses of 5/10mg/kg q2w
Drug: capecitabine [Xeloda] — Escalating doses of 500/650/750/900mg/m2 bid
Drug: erlotinib [Tarceva] — Escalating doses of 100/150mg daily

SUMMARY:
This 2 part study will evaluate the safety and efficacy of a combination of Avastin, Tarceva and Xeloda (ATX) as second-line treatment in patients with locally advanced and/or metastatic pancreatic cancer. In the first part of the study, cohorts of patients will receive escalating doses of combination treatment to determine the maximum tolerated dose. The recommended dose will be used in the second part of the study to determine the efficacy of the ATX regime, in terms of its effect on disease progression. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* pancreatic cancer with locally advanced and/or metastatic disease (stage IV);
* chemonaive for metastatic or locally advanced disease;
* ECOG performance status of 0-2.

Exclusion Criteria:

* local (stage IA to IIB)and locally advanced (stage III) pancreatic cancer;
* previous exposure to Avastin, Tarceva or Xeloda;
* other primary tumor within the last 5 years prior to enrollment, except for adequately treated cancer in situ of cervix, or basal cell skin cancer;
* current or recent chronic use of aspirin (>325 mg/day) or full therapeutic dose of anticoagulants or thrombolytic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty two (32) participants were included however, 2 participants discontinued before reaching the end of the evaluation period of 3 cycles of the complete study regimen (of all 3 drugs) at the recommended dose due to progressive disease.
Groups:
- ERL+BEV+CAP Dose Level-1: Participants were administered oral 100 milligrams (mg) of erlotinib (ERL) tablet daily at least 1 hour before or 2 hours after the ingestion of food, 5 milligrams per kilogram (mg/kg) of bevacizumab (BEV) intravenous (IV) infusion on Day 1 of each cycle (1 Cycle = 2 Weeks), and oral 500 milligrams per square meter (mg/m^2) of capecitabine (CAP) tablet twice daily (BID) within 30 minutes after the ingestion of food. All the medications were continued until confirmed evidence of disease progression or unacceptable toxicity.
- ERL+BEV+CAP Dose Level-2: Participants were administered oral 100 mg of erlotinib tablet daily at least 1 hour before or 2 hours after the ingestion of food, 5 mg/kg of bevacizumab IV infusion on Day 1 of each cycle (1 Cycle = 2 Weeks), and oral 650 mg/m^2 of capecitabine tablet BID within 30 minutes after the ingestion of food. All the medications were continued until confirmed evidence of disease progression or unacceptable toxicity.
- ERL+BEV+CAP Dose Level-3: Participants were administered oral 100 mg of erlotinib tablet daily at least 1 hour before or 2 hours after the ingestion of food, 5 mg/kg of bevacizumab IV infusion on Day 1 of each cycle (1 Cycle = 2 Weeks), and oral 800 mg/m^2 of capecitabine tablet BID within 30 minutes after the ingestion of food. All the medications were continued until confirmed evidence of disease progression or unacceptable toxicity.
- ERL+BEV+CAP Dose Level-4: Participants were administered oral 100 mg of erlotinib tablet daily at least 1 hour before or 2 hours after the ingestion of food, 5 mg/kg of bevacizumab IV infusion on Day 1 of each cycle (1 Cycle = 2 Weeks), and oral 900 mg/m^2 of capecitabine tablet BID within 30 minutes after the ingestion of food. All the medications were continued until confirmed evidence of disease progression or unacceptable toxicity.
- ERL+BEV+CAP Dose Level-5: Participants were administered oral 150 mg of erlotinib tablet daily at least 1 hour before or 2 hours after the ingestion of food, 5 mg/kg of bevacizumab IV infusion on Day 1 of each cycle (1 Cycle = 2 Weeks), and oral 800 mg/m^2 of capecitabine tablet BID within 30 minutes after the ingestion of food. All the medications were continued until confirmed evidence of disease progression or unacceptable toxicity.
- ERL+BEV+CAP Dose Level-6: Participants were administered oral 150 mg of erlotinib tablet daily at least 1 hour before or 2 hours after the ingestion of food, 10 mg/kg of bevacizumab IV infusion on Day 1 of each cycle (1 Cycle = 2 Weeks), and oral 800 mg/m^2 of capecitabine tablet BID within 30 minutes after the ingestion of food. All the medications were continued until confirmed evidence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | ERL+BEV+CAP Dose Level-1 | ERL+BEV+CAP Dose Level-2 | ERL+BEV+CAP Dose Level-3 | ERL+BEV+CAP Dose Level-4 | ERL+BEV+CAP Dose Level-5 | ERL+BEV+CAP Dose Level-6
Started | 6 | 6 | 6 | 6 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 6 | 3 | 3
Not completed — Major toxicity | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Disease progression | 4 | 5 | 3 | 4 | 2 | 3
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Missing documentation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — End of study visit not done | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Participant is unable to swallow drug | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Per-protocol population: All participants who received at least 1 evaluation period of 3 cycles of the complete study regimen (of all 3 drugs) at the recommended dose unless withdrawn from therapy earlier because of toxicity.
Groups:
- Triple Combination (Bevacizumab/Erlotinib/Capecitabine): Dose-escalation was performed using a substance-related toxicity-based dose escalation scheme and was started with capecitabine followed by erlotinib and completed by bevacizumab. Participants in different dose levels (Dose levels [DL]-1, 2, 3, 4, 5 and 6) were administered either oral 100 mg or 150 mg of erlotinib tablet daily, 5 mg/kg or 10 mg/kg of bevacizumab IV infusion on Day 1 of each cycle (1 Cycle = 2 Weeks), and any of the different doses of capecitabine BID (500/650/800/900 mg/m^2) orally. All the medications were continued until confirmed evidence of disease progression or unacceptable toxicity.
Arm/Group | Triple Combination (Bevacizumab/Erlotinib/Capecitabine)
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Maximum Tolerated Dose (MTD) of Capecitabine
Description: MTD for each of the medications was defined as the lowest dose studied which resulted in dose limiting toxicity (DLT) in at least 33 percent (%) of participants of the same quality category. DLT was defined as any greater than or equal to (>=) Grade (G) 3 or G4 toxicity; >= G3 non-hematological toxicities directly related to study treatment (other than untreated nausea/vomiting, alopecia, G3/G4 bilirubinemia for less than 7 days due to edema of the ductus choledochus and anemia); G4 thrombocytopenia, neutropenia lasting >= 7 days or G3 thrombocytopenia with complications, requiring transfusions, febrile neutropenia; stopping of oral CAP and/or ERL intake for >= 7 days, and/or cancellation of one or more BEV infusion(s) due to adverse events (AEs).
Time Frame: Up to Week 6 (Cycle 1-3)
Population: Per-protocol population.
Measure: Number; unit: mg/m^2 BID
Groups:
- Triple Combination (Bevacizumab/Erlotinib/Capecitabine): Dose-escalation was performed using a substance-related toxicity-based dose escalation scheme and was started with capecitabine followed by erlotinib and completed by bevacizumab. Participants in different dose levels (DLs - 1, 2, 3, 4, 5 and 6) were administered either 100 mg or 150 mg of erlotinib tablet orally daily, 5 mg/kg or 10 mg/kg of bevacizumab IV infusion on Day 1 of each cycle (1 Cycle = 2 Weeks), and any of the different doses of capecitabine BID (500/650/800/900 mg/m^2) orally. All the medications were continued until confirmed evidence of disease progression or unacceptable toxicity.
Arm/Group | Triple Combination (Bevacizumab/Erlotinib/Capecitabine)
Number analyzed (Participants) | 30
mg/m^2 BID | 900

2. Primary Outcome: Part 1: MTD of Erlotinib
Description: MTD for each of the medications was defined as the lowest dose studied which resulted in DLT in at least 33% of participants of the same quality category. DLT was defined as >= G3 or G4 toxicity; >= G3 non-hematological toxicities directly related to study treatment (other than untreated nausea/vomiting, alopecia, G3/G4 bilirubinemia for less than 7 days due to edema of the ductus choledochus and anemia); G4 thrombocytopenia, neutropenia lasting >= 7 days or G3 thrombocytopenia with complications, requiring transfusions, febrile neutropenia; stopping of oral CAP and/or ERL intake for >= 7 days, and/or cancellation of one or more BEV infusion(s) due to AEs.
Time Frame: Up to Week 6 (Cycle 1-3)
Population: Per-protocol population.
Measure: Number; unit: mg/day
Groups:
- Triple Combination (Bevacizumab/Erlotinib/Capecitabine): Dose-escalation was performed using a substance related toxicity-based dose escalation scheme and was started with capecitabine followed by erlotinib and completed by bevacizumab. Participants in different dose levels (DL-1, 2, 3, 4, 5 and 6) were administered with either 100 mg or 150 mg of erlotinib daily orally, 5 mg/kg or 10 mg/kg of bevacizumab IV infusion on Day 1 of each cycle (1 Cycle = 2 Weeks), and any of the different doses of capecitabine BID (500/650/800/900 mg/m^2) orally. All the medications were continued until confirmed evidence of disease progression or unacceptable toxicity.
Arm/Group | Triple Combination (Bevacizumab/Erlotinib/Capecitabine)
Number analyzed (Participants) | 30
mg/day | NA — DLTs were not observed for the maximum planned dose of erlotinib (150 mg/day) in the study; therefore, MTD was not defined for erlotinib.

3. Secondary Outcome: Part 1: Maximum Serum Concentration (Cmax) of Erlotinib and Its Metabolite OSI-420 (CP373420), Capecitabine and Its Metabolites (5'-Deoxy-5-Fluorocytidine [5'-DFCR] and 5'-Deoxy-5-Fluorouridine [5'-DFUR])
Time Frame: CAP: 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6 hours (h) of every 2-week cycle (until Week 259) ERL: 2, 3 4, 5, 6, 7, 8, 10, 24, 28, 48, 52, 72, 76, 96, 100, 120, 124, 144, 148, 168 and 172 h of every 2-week cycle (until Week 259)
Population: Per-protocol population. Here "n" signifies the number of participants who were evaluable for each drug for each arm, respectively.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (µg/mL)
Groups:
- ERL+BEV+CAP Dose Level-1: Participants were administered oral 100 mg of erlotinib tablet daily at least 1 hour before or 2 hours after the ingestion of food, 5 mg/kg of bevacizumab IV infusion on Day 1 of each cycle (1 Cycle = 2 Weeks), and oral 500 mg/m^2 of capecitabine tablet BID orally within 30 minutes after the ingestion of food. All the medications were continued until confirmed evidence of disease progression or unacceptable toxicity.
Arm/Group | ERL+BEV+CAP Dose Level-1 | ERL+BEV+CAP Dose Level-2 | ERL+BEV+CAP Dose Level-3 | ERL+BEV+CAP Dose Level-4 | ERL+BEV+CAP Dose Level-5 | ERL+BEV+CAP Dose Level-6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 3
micrograms per milliliter (µg/mL)
  Erlotinib (n=6,6,6,6,3,3) | 1.50 (1.21) | 0.95 (0.58) | 0.68 (0.34) | 0.93 (0.63) | 0.58 (0.15) | 1.69 (0.67)
  OSI-420 (n=6,6,6,6,3,3) | 0.09 (0.07) | 0.05 (0.03) | 0.04 (0.02) | 0.06 (0.04) | 0.03 (0.01) | 0.10 (0.02)
  Capecitabine (n=6,6,6,6,3,3) | 1.69 (1.22) | 1.13 (0.61) | 4.89 (4.23) | 5.48 (4.51) | 9.47 (5.19) | 9.9 (5.01)
  5'-DFCR (n=5,5,6,6,3,3) | 3.5 (3.02) | 4.28 (1.61) | 11.46 (5.32) | 6.26 (2.05) | 5.44 (2.43) | 4.15 (1.24)
  5'-DFUR (n=4,5,6,6,3,3) | 7.9 (4.41) | 7.3 (2.74) | 6.17 (2.63) | 7.24 (3.35) | 3.28 (0.72) | 5.1 (2.35)

4. Primary Outcome: Part 1: MTD of Bevacizumab
Description: as for outcome 2
Time Frame: Up to Week 6 (Cycle 1-3)
Population: Per-protocol population.
Measure: Number; unit: mg/kg once every 2 weeks (Q2W)
Arm/Group | Triple Combination (Bevacizumab/Erlotinib/Capecitabine)
Number analyzed (Participants) | 30
mg/kg once every 2 weeks (Q2W) | NA — DLTs were not observed for the maximum planned dose of bevacizumab (10 mg/kg once Q2W) in the study; therefore, MTD was not defined for capecitabine.

5. Primary Outcome: Part 1: Preliminary Recommended Dose (PRD) of Capecitabine for Part 2
Description: Once the MTD was reached then the preceding lower dose level was used as PRD. MTD for each of the medications was defined as the lowest dose studied which resulted in dose limiting toxicity (DLT) in at least 33% of participants of the same quality category. DLT was defined as >= G3 or G4 toxicity; >= G3 non-hematological toxicities directly related to study treatment (other than untreated nausea/vomiting, alopecia, G3/G4 bilirubinemia for less than 7 days due to edema of the ductus choledochus and anemia); G4 thrombocytopenia, neutropenia lasting >= 7 days or G3 thrombocytopenia with complications, requiring transfusions, febrile neutropenia; stopping of oral CAP and/or ERL intake for >= 7 days, and/or cancellation of one or more BEV infusion(s) due to AEs. If MTD was not defined for a drug treatment then the maximum planned dose of that particular drug was considered as PRD for Part 2.
Time Frame: Up to Week 6 (Cycle 1-3)
Population: Per-protocol population.
Measure: Number; unit: mg/m^2 BID
Arm/Group | Triple Combination (Bevacizumab/Erlotinib/Capecitabine)
Number analyzed (Participants) | 30
mg/m^2 BID | 800

6. Secondary Outcome: Part 1: Time to Reach Cmax (Tmax) of Erlotinib and Its Metabolite OSI-420 (CP373420), Capecitabine and Its Metabolites (5'-DFCR and 5'-DFUR)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hours (h)
Arm/Group | ERL+BEV+CAP Dose Level-1 | ERL+BEV+CAP Dose Level-2 | ERL+BEV+CAP Dose Level-3 | ERL+BEV+CAP Dose Level-4 | ERL+BEV+CAP Dose Level-5 | ERL+BEV+CAP Dose Level-6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 3
hours (h)
  Erlotinib (n=6,6,6,6,3,3) | 2.50 [1.00 to 8.00] | 2.00 [2.00 to 8.00] | 2.00 [1.00 to 6.00] | 3.00 [2.00 to 8.00] | 5.00 [4.00 to 6.00] | 2.00 [2.00 to 3.00]
  OSI-420 (n=6,6,6,6,3,3) | 3.00 [1.00 to 8.00] | 2.00 [2.00 to 24.00] | 2.00 [1.00 to 8.00] | 7.00 [2.00 to 24.00] | 6.00 [6.00 to 6.00] | 4.00 [2.00 to 4.00]
  Capecitabine (n=6,6,6,6,3,3) | 0.5 [0.5 to 5] | 1 [0.5 to 3] | 1.5 [0.5 to 3] | 0.75 [0.5 to 2] | 1 [0.5 to 2] | 0.5 [0.5 to 1]
  5'-DFCR (n=5,5,6,6,3,3) | 0.5 [0.5 to 2.5] | 1 [1 to 1.5] | 1.5 [0.5 to 2.5] | 1 [0.5 to 2] | 1 [0.5 to 2.5] | 1.5 [0.5 to 2.5]
  5'-DFUR (n=4,5,6,6,3,3) | 1 [1 to 2.5] | 1.5 [1 to 2] | 1.5 [0.5 to 2.5] | 1.5 [0.5 to 2] | 1 [0.5 to 2.5] | 1.5 [1 to 2]

7. Secondary Outcome: Part 1: Last Quantifiable Drug Concentration (Clast) of Erlotinib and Its Metabolite OSI-420 (CP373420), Capecitabine and Its Metabolites (5'-DFCR and 5'-DFUR)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | ERL+BEV+CAP Dose Level-1 | ERL+BEV+CAP Dose Level-2 | ERL+BEV+CAP Dose Level-3 | ERL+BEV+CAP Dose Level-4 | ERL+BEV+CAP Dose Level-5 | ERL+BEV+CAP Dose Level-6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 3
µg/mL
  Erlotinib (n=6,6,6,6,3,3) | 0.37 (0.36) | 0.31 (0.19) | 0.23 (0.11) | 0.39 (0.39) | 0.23 (0.02) | 0.52 (0.19)
  OSI-420 (n=6,6,6,6,3,3) | 0.04 (0.06) | 0.02 (0.01) | 0.01 (0.01) | 0.04 (0.04) | 0.01 (0.00) | 0.04 (0.01)
  Capecitabine (n=6,6,6,6,3,3) | 0.05 (0.06) | 0.2 (0.2) | 0.17 (0.15) | 0.06 (0.03) | 0.29 (0.26) | 0.17 (0.1)
  5'-DFCR (n=5,5,6,6,3,3) | 0.23 (0.23) | 0.08 (0.04) | 0.64 (0.6) | 0.75 (0.89) | 0.99 (1.22) | 0.3 (0.1)
  5'-DFUR (n=4,5,6,6,3,3) | 2.54 (0.14) | 1.03 (1.05) | 0.77 (0.92) | 0.58 (0.49) | 0.14 (0.08) | 0.14 (0.05)

8. Secondary Outcome: Part 1: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Measurable Concentration (AUClast) of Erlotinib and Its Metabolite OSI-420 (CP373420), Capecitabine and Its Metabolites (5'-DFCR and 5'-DFUR)
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*µg/mL
Arm/Group | ERL+BEV+CAP Dose Level-1 | ERL+BEV+CAP Dose Level-2 | ERL+BEV+CAP Dose Level-3 | ERL+BEV+CAP Dose Level-4 | ERL+BEV+CAP Dose Level-5 | ERL+BEV+CAP Dose Level-6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 3
h*µg/mL
  Erlotinib (n=6,6,6,6,3,3) | 15.81 (12.91) | 11.06 (5.41) | 9.15 (4.39) | 13.07 (11.03) | 8.54 (1.96) | 19.88 (4.75)
  OSI-420 (n=6,6,6,6,3,3) | 1.15 (1.21) | 0.48 (0.35) | 0.41 (0.18) | 0.99 (0.73) | 0.36 (0.03) | 1.42 (0.17)
  Capecitabine (n=6,6,6,6,3,3) | 1.43 (1.02) | 1.63 (1.01) | 5.88 (6.28) | 5.28 (3.25) | 13.63 (8.63) | 9.74 (3.02)
  5'-DFCR (n=5,5,6,6,3,3) | 3.97 (2.65) | 7.01 (1.89) | 20.27 (11.53) | 9.35 (3.26) | 12.63 (9.89) | 8.06 (2.14)
  5'-DFUR (n=4,5,6,6,3,3) | 15.42 (9.45) | 13.58 (7.84) | 9.76 (4.60) | 10.86 (4.96) | 5.17 (0.89) | 8.53 (1.87)

9. Secondary Outcome: Part 2: Percentage of Participants Free From Disease Progression
Description: As per Response Evaluation Criteria In Solid Tumors (RECIST) version (v) 1.1, progressive disease (PD) is defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of 1 or more new lesions (target and non-target lesions) or the unequivocal progression of existing non-target lesions.
Time Frame: Month 6
Population: Data was not reported as there were no participants analyzed since Part 2 of the study was not fully implemented.
Arm/Group | ERL+BEV+CAP Dose Level-1 | ERL+BEV+CAP Dose Level-2 | ERL+BEV+CAP Dose Level-3 | ERL+BEV+CAP Dose Level-4 | ERL+BEV+CAP Dose Level-5 | ERL+BEV+CAP Dose Level-6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Part 2: Percentage of Participants With Disease Control
Description: A participant was defined as having controlled disease if they sustained a Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) during the assessment. As per RECIST v1.1, CR is defined as the disappearance of all target and non-target lesions and normalization of tumor marker level; PR is defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the screening sum longest diameter; SD for target lesions is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the treatment started and SD for non-target lesions defined as persistence of 1 or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits.
Time Frame: From baseline thereafter, every 6 weeks (±7 days), then 1 week after last dose (follow-up), thereafter every 6 weeks (±7 days) until disease progression (up to Week 259)
Population: Data was not reported as there were no participants analyzed since Part 2 of the study was not fully implemented.
Arm/Group | ERL+BEV+CAP Dose Level-1 | ERL+BEV+CAP Dose Level-2 | ERL+BEV+CAP Dose Level-3 | ERL+BEV+CAP Dose Level-4 | ERL+BEV+CAP Dose Level-5 | ERL+BEV+CAP Dose Level-6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Part 2: Percentage of Participants With Clinical Benefit Response
Description: Clinical benefit response was defined as a composite of pain control, Karnofsky performance status (KPS), and weight. The KPS allows participants to be classified as per their functional impairment (abnormal function). It was recorded on an 11-point scale; 0= "dead" to 100= "Normal, no complaints, no evidence of disease" and sub-divided to 3 categories; 0 to 40 = "Unable to care for self, requires institutional or hospital care or equivalent, disease may be rapidly progressing"; 50 to 70= "Unable to work, able to live at home and care for most personal needs, varying amount of assistance needed and 80 to 100= "Able to carry on normal activity; no special care is needed".
Time Frame: One week before start of study treatment and weekly until disease progression or death (Up to Week 259)
Population: Data was not reported as there were no participants analyzed since Part 2 of the study was not fully implemented.
Arm/Group | ERL+BEV+CAP Dose Level-1 | ERL+BEV+CAP Dose Level-2 | ERL+BEV+CAP Dose Level-3 | ERL+BEV+CAP Dose Level-4 | ERL+BEV+CAP Dose Level-5 | ERL+BEV+CAP Dose Level-6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Part 2: Overall Survival
Description: Survival was the interval of time from date of first dose of study medication to date of death at any time. Participants who had not died were censored at the date of last contact when they were known to be alive.
Time Frame: From baseline until death (Up to Week 259)
Population: Data was not reported as there were no participants analyzed since Part 2 of the study was not fully implemented.
Arm/Group | ERL+BEV+CAP Dose Level-1 | ERL+BEV+CAP Dose Level-2 | ERL+BEV+CAP Dose Level-3 | ERL+BEV+CAP Dose Level-4 | ERL+BEV+CAP Dose Level-5 | ERL+BEV+CAP Dose Level-6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Part 1: PRD of Erlotinib for Part 2
Description: Once the MTD was reached then the preceding lower dose level was used as PRD. MTD for each of the medications was defined as the lowest dose studied which resulted in DLT in at least 33% of participants of the same quality category. DLT was defined as >= G3 or G4 toxicity; >= G3 non-hematological toxicities directly related to study treatment (other than untreated nausea/vomiting, alopecia, G3/G4 bilirubinemia for less than 7 days due to edema of the ductus choledochus and anemia); G4 thrombocytopenia, neutropenia lasting >= 7 days or G3 thrombocytopenia with complications, requiring transfusions, febrile neutropenia; stopping of oral CAP and/or ERL intake for >= 7 days, and/or cancellation of one or more BEV infusion(s) due to AEs. If MTD was not defined for a drug treatment then the maximum planned dose of that particular drug was considered as PRD for Part 2.
Time Frame: Up to Week 6 (Cycle 1-3)
Population: Per-protocol population.
Measure: Number; unit: mg/day
Arm/Group | Triple Combination (Bevacizumab/Erlotinib/Capecitabine)
Number analyzed (Participants) | 30
mg/day | 150

14. Primary Outcome: Part 1: PRD of Bevacizumab for Part 2
Description: as for outcome 13
Time Frame: Up to Week 6 (Cycle 1-3)
Population: Per-protocol population.
Measure: Number; unit: mg/kg Q2W
Arm/Group | Triple Combination (Bevacizumab/Erlotinib/Capecitabine)
Number analyzed (Participants) | 30
mg/kg Q2W | 10

ADVERSE EVENTS:
Time Frame: From screening up to 30 days after the last chemotherapy treatment.
Groups:
- ERL+BEV+CAP Dose Level-1: Participants were administered oral 100 mg of erlotinib tablet daily at least 1 hour before or 2 hours after the ingestion of food, 5 mg/kg of bevacizumab IV infusion on Day 1 of each cycle (1 Cycle = 2 Weeks), and oral 500 mg/m^2 of capecitabine tablet BID within 30 minutes after the ingestion of food. All the medications were continued until confirmed evidence of disease progression or unacceptable toxicity.
Arm/Group | ERL+BEV+CAP Dose Level-1 | ERL+BEV+CAP Dose Level-2 | ERL+BEV+CAP Dose Level-3 | ERL+BEV+CAP Dose Level-4 | ERL+BEV+CAP Dose Level-5 | ERL+BEV+CAP Dose Level-6
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/6 | 4/6 | 5/6 | 3/3 | 3/3
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 6/6 | 6/6 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ERL+BEV+CAP Dose Level-1 (N=6) | ERL+BEV+CAP Dose Level-2 (N=6) | ERL+BEV+CAP Dose Level-3 (N=6) | ERL+BEV+CAP Dose Level-4 (N=6) | ERL+BEV+CAP Dose Level-5 (N=3) | ERL+BEV+CAP Dose Level-6 (N=3)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bilirubinaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Embolism pulmonary (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyponatremia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage rectum (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fever (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Skeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ERL+BEV+CAP Dose Level-1 (N=6) | ERL+BEV+CAP Dose Level-2 (N=6) | ERL+BEV+CAP Dose Level-3 (N=6) | ERL+BEV+CAP Dose Level-4 (N=6) | ERL+BEV+CAP Dose Level-5 (N=3) | ERL+BEV+CAP Dose Level-6 (N=3)
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 3 | 1 | 1
Bilirubin (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1 | 0 | 0
Coagulation time decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Blood and lymphatic system disorders) | 1 | 1 | 3 | 1 | 0 | 0
Gingival bleeding (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1 | 0 | 0
Hypoproteinemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 3 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 3 | 2 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 4 | 4 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 0 | 0
Gastrointestinal disorder nos (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0
Hematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hiccup (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Melena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mouth dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 2 | 4 | 4 | 2 | 2
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 4 | 4 | 1 | 1
Back pain (General disorders) | 1 | 1 | 1 | 0 | 0 | 0
Common cold (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
Exsiccosis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 6 | 3 | 3 | 3 | 2 | 2
Fever (General disorders) | 0 | 2 | 0 | 1 | 0 | 0
Leg pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Oedema mouth (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 0 | 1 | 2 | 0 | 0
Pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Rigors (General disorders) | 0 | 0 | 0 | 2 | 1 | 0
Syncope (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Temperature changed sensation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0
Moniliasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Wound dehiscence (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
C- reactive protein positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Appetite loss (Metabolism and nutrition disorders) | 4 | 1 | 2 | 4 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Weight decrease (Metabolism and nutrition disorders) | 1 | 0 | 2 | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Skeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Dysphonia (Nervous system disorders) | 1 | 0 | 2 | 2 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Taste perversion (Nervous system disorders) | 1 | 1 | 2 | 1 | 0 | 1
Vertigo (Nervous system disorders) | 1 | 1 | 1 | 1 | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 2 | 0 | 0 | 0
Albuminuria (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 1 | 1
Genital ulceration (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vaginitis (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 0 | 1
Increased pulmonary secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1 | 0 | 0
Bullous eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mucosis left breast (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodyesthesia (Skin and subcutaneous tissue disorders) | 2 | 5 | 3 | 3 | 1 | 0
Paronychia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 | 5 | 4 | 4 | 2 | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin dry (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 2 | 1 | 0
Skin reaction localized (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sweating increased (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1 | 2 | 0 | 1
Hypertension aggravated (Vascular disorders) | 2 | 1 | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
(Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Planned Part 2 of the study was not implemented and outcome measures related to Part 2 were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.